CLINICAL TRIAL: NCT04954404
Title: Transcatheter Mitral Valve InterventiOn Single Center Registry in CHinese Patients With Mitral Valve Disease (TORCH-M)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0593
Record Dates: First submitted 2021-06-20; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Intervention Model Description: Transcatheter mitral valve repair/Transcatheter mitral valve replacement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter mitral valve repair/replacement (Experimental)
  Interventions: Device: transcatheter mitral valve repair/transcatheter mitral valve replacement

INTERVENTIONS:
Device: transcatheter mitral valve repair/transcatheter mitral valve replacement — transcatheter mitral valve repair/transcatheter mitral valve replacement

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of transcatheter mitral valve intervention in Chinese population with mitral valve disease.

DETAILED DESCRIPTION:
Prospective, single-arm, single-center clinical evaluation of transcatheter mitral valve intervention in subjects with mitral valve disease who are treated per standard of care and who have been determined by the local heart team as appropriate for interventional treatment. Eligible subjects will be treated by transcatheter mitral valve repair or transcatheter mitral valve replacement.

This single-arm registry will provide valuable new information regarding use of multiple mitral valve interventional devices and evaluate the safety and effectiveness of transcatheter mitral valve intervention in Chinese population with mitral valve disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mitral valve disease, as determined by the site from a transthoracic echocardiogram (TTE), and in the judgment of the investigator intervention is likely to provide clinical benefit for the patient.
2. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
3. The subject agrees to comply with specified follow-up evaluations and to return to the investigational site where the procedure was performed.
4. Patients are technical and anatomical eligible for interventions.

Exclusion Criteria:

1. In the judgment of the investigator, subjects are not anatomical eligible for interventions.
2. Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically.
3. Active endocarditis or active rheumatic heart disease.
4. History of severe bleeding diathesis or coagulopathy or subject will refuse blood transfusions.
5. Subject has any kind of conditions that might prevent patients benefiting from therapeutic benefit (i.e., Severe mental illness) or life expectancy is less than one year.
6. Subject has any kind of disorder per investigator's judgement that compromises his/her ability to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes of all-cause mortality and rate of rehospitalization related to heart failure. | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Composite outcomes of all-cause mortality and rate of rehospitalization related to heart failure.

SECONDARY OUTCOMES:
All-cause mortality | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Death from any causes including both cardiovascular and non-cardiovascular.
Cardiovascular mortality | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Death from any cardiovascular events.
Rehospitalization related to heart failure | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Number of patients readmission for recurrent Heart Failure.
Stroke | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Transient ischemic attack | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Brain lesion | Predischarge
  Number and volumes of new brain lesions detected by Magnetic Resonance Imaging (MRI) after procedure with or without clinical symptom.
Myocardial infarction | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Vascular complications | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Bleeding events | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Permanent pacemaker implantation | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Device success | Immediately after procedure
  Defined according to consensus document from the mitral valve academic research consortium (MVARC).
Infective endocarditis | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Number of patients with infective endocarditis.
Recurrent hospitalization - All cause | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Number of patients hospitalized for≥24h. Hospitalizations planned for pre-existing conditions are excluded unless there is worsening of the baseline condition according to MVARC.
Acute kidney injury | Predischarge, 30 days
New-onset atrial fibrillation | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Change of New York Heart Association functional classification | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Change of NYHA status from baseline to each follow-up.
MR and/or MS severity | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  The change in MR and/or MS severity from baseline to each follow-up.
Quality of life improvement | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Improvement in quality of life from baseline to each follow-up measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Modified Rankin scale score | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Change of cognitive function | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Change of cognitive function from baseline to each follow-up measured by the Mini-mental State Examination （MMSE）.
6-min walk test | 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  The change in 6-min walk test distance from baseline to each follow-up.
Reintervention of mitral valve | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Any conditions need reintervention or surgery, as device-related thrombosis, valve deterioration.
Significant iatrogenic atrial septal defect | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
  Number of patients reported as clinically significant iASD requiring ASD closure.
Device embolization or single leaflet device attachment | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Effective regurgitant orifice area | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Regurgitant volume | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Regurgitant fraction | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Mitral valve area | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Mean mitral valve gradient | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Left ventricular ejection fraction (LVEF) | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Left ventricular end-diastolic diameter (LVEDD) | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Left ventricular end-systolic diameter (LVESD) | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Pulmonary artery systolic pressure (PASP) | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Right ventricular systolic pressure (RVSP) | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
Left ventricular mass | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years
BNP and/or NT-proBNP levels | Predischarge, 30 days, 6 months, 1 year, 2 years, 3 years, 5 years, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, PhD, MD, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine., Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Pu Z, Yu T, Liu X, Lin X, Li H, Lim DS, Wang J. A modified Carpentier classification in transcatheter edge-to-edge repair for mitral regurgitation. Catheter Cardiovasc Interv. 2024 Oct;104(4):870-877. doi: 10.1002/ccd.31158. Epub 2024 Jul 24. PMID 39049480